CLINICAL TRIAL: NCT05799885
Title: The Effects of Combined Neuro-vestibular-ocular Exercises and Myofascial Release on Proprioception and Performance in Soccer Players With Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: YEDITEPEU-BUSRAKOCAKILIC-0096
Record Dates: First submitted 2023-02-13; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-01

CONDITIONS: Ankle Inversion Sprain; Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 31 players with ankle instability (Experimental): 2 sessions per week for 8 weeks, total training time 30 min
  Interventions: Other: Myofascial Release group
- 30 players with ankle instability (Experimental): 2 sessions per week for 8 weeks, total training time 30-40 min
  Interventions: Other: Neuro-vestibular-ocular group

INTERVENTIONS:
Other: Neuro-vestibular-ocular group — Neuro-vestibular-ocular exercise group (30 footballers)will do the exercises given in addition to their training
  Arms: 30 players with ankle instability
Other: Myofascial Release group — Manual myofascial release will be applied by the physiotherapist.(30 football players)
  Arms: 31 players with ankle instability

SUMMARY:
Chronic ankle instability was first defined by Freeman as recurrent ankle sprains following an ankle sprain and the feeling of dislocation in the ankle lasting longer than six months. The recurrence of ankle sprains in athletes leads to the realization of ankle instability. Functional ankle instability gives the feeling that a re-sprain will occur at any time due to decreased static and dynamic support in the joint.Neuro-vestibular-ocular exercises is an approach that combines neuromuscular training and vestibular-ocular training techniques.At the same time, we are doing this study because of the mixed studies on the effect of fascial relaxation on the performance and proprioception of a specific group of football players.

DETAILED DESCRIPTION:
A total of 60 football players with instability <27 according to the CAIT scale, whose proprioception and performance (jump, sprint, zig-zag test, kick speed) values were taken at the beginning, will be divided into two groups.Myofascial release will be applied to the lower extremity posterior line chain described by Myers by the physiotherapist to the first group.The other group (30 people) will be given neuro-vestibular-ocular exercises.Both groups will continue their training programme as ready.The training will be done in 2 sessions and 30 minutes per week.

ELIGIBILITY:
Inclusion Criteria:

* a history of 'giving way' and/or recurrent sprains and/or 'feeling of instability' in the injured ankle joint within the last 6 months.
* decreased function due to ankle sprain history
* "feeling of instability" will be defined as ≤27 points on the Cumberland ankle instability scale (CAIT) and the most affected side will be determined as the relevant limb for testing. CAIT score between right and left foot The dominant ankle will be selected.
* Having had at least two previous lateral sprains in the same ankle.

Exclusion Criteria:

* history of musculoskeletal surgery and/or fractures in the lower extremities;
* acute injury to the musculoskeletal structures of other lower extremity joints in the last three months that affects joint integrity and function and causes interruption of desired physical activity for at least one day;
* having a history of balance and vestibular disorders.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-04-02 (Estimated); Primary Completion 2023-09-03 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
CAIT Scale | a day before the rehabilitation-at the time of discharge(8 weeks)
  Participants will be included based on the CAIT questionnaire and who get 27 points or less from this questionnaire. In the test, cut off score of less or equal to 27 as indicate of chronic ankle instability. The precision of the instrument is increased as it is a multiple answer option instrument. The CAIT is able to measure the severity of instability by using a numeric value and also can be filled out for both the left and right ankle, making it possible to assess both ankles individually.

SECONDARY OUTCOMES:
proprioception evaluation | a day before the rehabilitation-at the time of discharge(8 weeks)
  The goniometer is used as a tool to measure proprioceptive perception of the ankle joint.
  Subjects are placed in the starting position with their eyes closed. The ankle subtalar joint is in neutral position (STJN) and the goniometer is set to zero. 20 degrees of inversion and 10 degrees of eversion are passively performed on the ankle and it is placed in neutral position.(13) The measurements are repeated 3 times and deviations from the target angle are measured with a goniometer.
Landing Error Scoring System (LESS) | a day before the rehabilitation-at the time of discharge(8 weeks)
  Jumping performance will be measured by Landing Error Scoring System (LESS). Materials required for this;12 inch platform Target line (At a distance of half the subjects height)2 cameras at 1 meter height (At 10 feet in front of the landing area and at 10 feet to the right of the landing area)LESS scale.The athlete is instructed to jump forward from the box with both feet.Both feet should make contact beyond the target line.After contact, jump right back up to maximal height and land again on both feet.This is repeated for three trials.The video of the jumps is taken from both the cameras in front and at the side.The feet, ankle, knees, hip, trunk, shoulder, neck and head posture is assessed through the video.It is a 19-point continuous scale. According to the performance sheet, the questions 1-15 are Yes/No questions that are rated as 0 or 1. The questions 16 and 17 are rated as 0,1 and 2 depending on the joint displacement
30 meters Sprint Test | a day before the rehabilitation-at the time of discharge(8 weeks)
  Sprint performance will be assessed by a 30-meter sprint test. A maximal 30 m sprint will be performed 3 times on the field. There is a 3-minute recovery period between the 30-m sprints. The shortest time taken to cover the 30 m distance in the sprint test will be taken into account.
Zigzag agility test(with and without the ball) | a day before the rehabilitation-at the time of discharge(8 weeks)
  There was a recovery time of 2 minutes between trials. The shortest time will be recorded as the performance of the zigzag agility tests with and without the ball. In the test, 4 cones are placed at the corners and 1 cone is placed in the center of the track. The long side of the track is 4,05 m (16 feet), the short side is 3 m (10 feet) (1feet=0,3 m)In the zigzag agility test with the ball, there is no specific rule such as the number of ball contacts. Time was measured using a stopwatch
Kick Speed | a day before the rehabilitation-at the time of discharge(8 weeks)
  The ball will be placed 11 meters away from the goal line. Cones will be placed 1 and 2 meters away from the starting position of the ball. The player will stand next to the cone at the 2nd meter and accelerate. Participants will be asked to kick the ball as fast as possible using the inside of the unstable foot. The measurement will be done with the apple app called "speed gun". The rest time between attempts will be 20 seconds. They will be told not to reduce the speed to improve the accuracy of the shot, the best time will be included in the trial results.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kocakılıç, master, Principal Investigator — Yeditepe University
Locations (1):
- Büşra, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No